CLINICAL TRIAL: NCT03247257
Title: Epidural Versus General Anesthesia for Laparoendoscopic Single Site Cholecystectomy: A Prospective, Comparative, Controlled, Blinded Study
Brief Title: Comparing Epidural Versus General Anesthesia for LESS Cholecystectomies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Florida Hospital Tampa Bay Division (Other)
Responsible Party: Principal Investigator, Alexander Rosemurgy, Director Surgical Digestive Disorders and GERD Center, Florida Hospital Tampa Bay Division
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 482717 revised
Record Dates: First submitted 2017-07-26; First posted 2017-08-11 (Actual); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Cholelithiasis
MeSH Terms: conditions — Cholelithiasis | interventions — Anesthesia, General; Propofol; Anesthesia, Epidural

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: General Anesthesia (Active Comparator): 35 patients will be randomized to receive general anesthesia during their laparoendoscopic single site incision cholecystectomy.
  Interventions: Procedure: General Anesthesia
- Group B: Epidural Anesthesia (Active Comparator): 35 patients will be randomized to receive epidural anesthesia during their laparoendoscopic single site incision cholecystectomy.
  Interventions: Procedure: Epidural Anesthesia

INTERVENTIONS:
Procedure: General Anesthesia — Patients will be put under general anesthesia for cholecystectomy
  Other Names: IV propofol
  Arms: Group A: General Anesthesia
Procedure: Epidural Anesthesia — Patients will receive Epidural Anesthesia for cholecystectomy
  Other Names: Epidural lidocaine
  Arms: Group B: Epidural Anesthesia

SUMMARY:
This study is a prospective, comparative, controlled, blinded study that will enroll a total of 70 adults that will undergo elective laparoendoscopic single-site incision gallbladder removal. The objective of this study is to compare Epidural versus General Anesthesia for postoperative pain, length of hospital stay, outcomes, and cost of post-cholecystectomy patients.

DETAILED DESCRIPTION:
This is a prospective, comparative, controlled, blinded study that will enroll a total of 70 adult patients that require an elective cholecystectomy.

Patients will be randomized 1:1 to receive either general anesthesia (Group A) or epidural anesthesia (Group B) for their laparoendoscopic single site incision (LESS) gallbladder removal surgery (cholecystectomy). Randomization will be achieved using a computer-generated list. The patient will know what are they are randomized to before entering the operating room because an epidural will need to be placed preoperatively. Standards for basic anesthetic monitoring approved by the American Society of Anesthesiologists will occur intraoperatively.

Postoperative evaluations will be completed by a medical professional that is blinded to the type of anesthesia used during the LESS surgery. Postoperative evaluations include a physical exam, adverse events, medication administration, vital signs and post-anesthesia recovery score for ambulatory patients (PARSAP) scores will be taken every 15 minutes until the patient has a score of at least 18.

Patients will be followed 90 days postoperatively to collect pain scores, analgesic use, adverse events, and quality of life questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 65 years of age
* ASA I or II
* Patient has a diagnosis of biliary colic with documented cholecystitis, symptomatic gallstones, polyps by imaging or biliary dyskinesia with documented EF < 30%
* No cardiopulmonary disease
* Normal coagulation profile

Exclusion Criteria:

* Any female patient, who is pregnant, suspected pregnant, or nursing
* Contraindication for pneumoperitoneum
* Contraindication for epidural anesthesia
* Allergy to local anesthetic agents
* Any patient with acute calculus or acalculous cholecystitis
* Any patient who has had an upper midline or right sub costal incision
* Any patient with preoperative indication for a cholangiogram
* Any patient with ASA ≥ 3
* Any patient who is undergoing Peritoneal Dialysis (PD)
* History of long term analgesic use requiring pain management (>1 week)
* Any patient who has an unrepaired umbilical hernia or has had prior umbilical hernia repair
* Any patient with obstructive sleep apnea (OSA), history of OSA or at high risk of OSA as determined by the STOP Questionnaire
* BMI > 35 kg/m2
* Any patient with a history of severe, uncontrolled GERD

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-02; Primary Completion 2018-12 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Post Anesthesia Recovery Score for Ambulatory Patients | Immediately postoperative
  PARSAP scores in the post-anesthesia recovery unit

SECONDARY OUTCOMES:
SF-12 Health survey scores | Postoperative days 1, 6, 7/8/9 or 10, 30, 90
  scale of 12-47
Pain | Immediately postoperative through postoperative day 90
  VAS 0-10 scale
Opioid requirement | Preoperative through postoperative day 90
  Opioid use in milligrams through postoperative day 90 will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Sharona Ross, MD, Principal Investigator — Florida Hospital Tampa; Alexander Rosemurgy, MD, Principal Investigator — Florida Hospital Tampa
Locations (1):
- Florida Hospital Tampa, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided